CLINICAL TRIAL: NCT05600712
Title: A Retro/Prospective Multi-Centre Data Capture on REDAPT Sleeved Stem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FORESN2
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Safety and Performance

STUDY DESIGN:
Intervention Model Description: Participants who have been implanted with REDAPT Sleeved Stem
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- single arm (Other): subjects who have redapt sleeved stem implant
  Interventions: Device: REDAPT Sleeved Stem

INTERVENTIONS:
Device: REDAPT Sleeved Stem — The REDAPT Sleeved Stem is designed to provide secondary proximal support to the distal fixation and enhance implant stability.

SUMMARY:
Retro/Prospective study to collect 2 year follow-up on REDAPT sleeved stem.

DETAILED DESCRIPTION:
The purpose of this study is to assess performance and safety of the Smith & Nephew REDAPT Sleeved Stem by collecting retrospective 2 year post-op with PROMs or prospective 2 year post-op with PROMs.

ELIGIBILITY:
Inclusion Criteria:

* Primary and revision surgery for hip degenerative joint disease including osteoarthritis, avascular necrosis, and traumatic arthritis.
* Rheumatoid arthritis, congenital dysplasia, femoral neck fracture, trochanteric fractures of the proximal femur with head involvement, and fracture-dislocation of the hip.

Exclusion Criteria:

* Conditions that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriate size implant (blood supply limitations, osteoporosis/metabolic disorders, infections)
* Mental or neurological conditions impairing or precluding cooperation with post-operative protocols and proper response to PROMs.
* Skeletal immaturity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Harris HIp Score (HHS) | 2 years
  measures pain, function, absence of deformity and range of motion after hip surgery. This is performed by a qualified health care provider. The higher the score, the better the outcome.
Hip Disablity and Osterarthritis Outcome Score (HOOS) | 2 year
  Scoring from 0-100 with 0 indicating the worst possible hip symptoms and 100 indicating no symptoms. This tool assesses patients opinion of their hip and associated problems, evaluate symptoms and functional limitations. There are 40 items assessing 5 subscales of: Pain, symptoms, activities of daily living (ADL), function in sport and recreation and Hip related quality of life.
HOOS Jr. | 2 year
  Scoring from 0-100 with 0 indicating the worst possible hip symptoms and 100 indicating no symptoms. This tool assesses patients opinion of their hip and associated problems, evaluate symptoms and functional limitations. this version is shortened to 6 questions assessing function, pain and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation for Orthopaedic Research and Education, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No